CLINICAL TRIAL: NCT00278486
Title: Immune Ablation and Hematopoietic Stem Cell Transplantation in Patients With Autoimmune-Related Retinopathy and Optic Neuropathy (ARRON) Syndrome (Not Associated With Cancer)
Brief Title: Hematopoietic Stem Cell Transplantation in Autoimmune-Related Retinopathy(ARRON)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: First subject over five years after the transplant. The second subject is not in compliance with follow ups. We do not plan to enroll more subjects.
Sponsor: Richard Burt, MD (Other)
Responsible Party: Sponsor-Investigator, Richard Burt, MD, MD, Northwestern University
Organization: Northwestern University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DI ARRON 04
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stem cell transplantation (Experimental)
  Interventions: Biological: Hematopoietic stem cell transplantation.

INTERVENTIONS:
Biological: Hematopoietic stem cell transplantation. — Autologous hematopoietic stem cell transplantation will be performed.

SUMMARY:
ARRON is a disease believed to be due to immune cells, cells which normally protect the body, but are now attacking the tissue in the retina and/or optic nerve. In addition, the disease may affect the nerves in the ear or other parts of the body . The affected nerves fail to respond, or respond only weakly, to stimuli causing numbing, tingling, pain, and progressive muscle weakness. If the nerves to the ear are affected, reduced hearing or deafness may result. The likelihood of progression of your disease is high. This study is designed to examine whether treating patients with high dose cyclophosphamide and rabbit ATG (drugs which reduce the function of the immune system) followed by return of previously collected blood stem cells will stop the progression of ARRON syndrome. Stem cells are undeveloped cells that have the capacity to grow into mature blood cells, which normally circulate in the blood stream. The purpose of the cyclophosphamide and rabbit ATG is to destroy the cells in the immune system which are thought to be causing this disease. The purpose of the stem cell infusion is to restore the body's blood production, which will be severely impaired by the high dose chemotherapy and to produce a normal immune system that will no longer attack the body.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-60.
2. Diagnosis of ARRON syndrome. Diagnostic criteria described below.

   Unexplained visual loss over weeks to months. The visual loss includes both visual acuity and field loss define as follows:
   * Visual acuity: 20/40 or less

   OR
   * Visual field: perimetric mean deviation -5b

     * Positive antibody to retina or optic nerve.

   OR

   A response to immunosuppressive drugs or immune modulators (response is defined by improvement of vision or decrease the rate of decline of visual loss).
   * Absence of malignancy {negative physical examination, gastrointestinal endoscopies, mammography and gynecologic examination (for female), and serum PSA measurement (for male) within a year}.
   * Negative MRI of brain.
3. The patient has failed at least 3 months of corticosteroids (prednisone 0.5mg/kg to start), IVIG and at least one other immunosuppressive drug such as methotrexate, Imuran, cyclosporine, etc. Failure is defined by decline of visual acuity (by standard Snellen acuity clinical testing) or visual field (by Humphrey Automated Machine with the 30-2 program or using Kinetic Visual Fields on the Goldman Perimeter)

Exclusion Criteria:

1. Absence of light perception lasting more than 6 months
2. Any illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy.
3. Prior history of malignancy except localized basal cell, squamous skin cancer or carcinoma in situ of the cervix. Other malignancies for which the patient is judged to be cured, such as head and neck cancer, or breast cancer will be considered on an individual basis.
4. Positive pregnancy test.
5. Inability or unwillingness to pursue effective means of birth control. Effective birth control is defined as 1) refraining from all acts of vaginal intercourse (ABSTINENCE); 2) consistent use of birth control pills; 3) injectable birth control methods (Depo-provera, Norplant); 4) tubal sterilization or male partner who has undergone vasectomy; 5) placement of an IUD (intrauterine device); or 6) use, with every act of intercourse, of diaphragm with contraceptive jelly and/or condoms with contraceptive foam.
6. Failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
7. FEV1/FVC < 60% of predicted after bronchodilator therapy (if necessary).
8. DLCO < 50% of predicted.
9. Active ischemic heart disease and/or those who have had a myocardial infarction within 6 months.
10. Resting LVEF < 40 %.
11. Bilirubin > 2.0 mg/dl
12. Serum creatinine > 2.0 mg/dl.
13. Known hypersensitivity to mouse, rabbit, or E. Coli derived proteins, or to iron compounds/medications.
14. Presence of metallic objects implanted in the body that would preclude the ability of the patient to safely have MRI exams.
15. Diagnosis of primary progressive MS.
16. Platelet count < 100,00/ul
17. Psychiatric illness, mental deficiency or cognitive dysfunction making compliance with treatment or informed consent impossible.
18. Active infection except asymptomatic bacteruria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2004-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Standard Snellen acuity clinical testing and improvement visual fields is done by using Humphrey Automated Machine with 30-2 program or using Kinetic Visual Fields on the Goldman Perimeter) | 5 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States